CLINICAL TRIAL: NCT00014521
Title: Phase I Evaluation Of The Safety Of Karenitecin In The Treatment Of Recurrent Malignant Gliomas
Brief Title: Karenitecin in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068552; NABTT-2006; JHOC-NABTT-2006
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2005-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Gliosarcoma | interventions — cositecan

INTERVENTIONS:
Drug: karenitecin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of karenitecin in treating patients who have recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of karenitecin in patients with recurrent malignant glioma who are receiving or not receiving anticonvulsants known to be metabolized by the P450 hepatic enzyme complex.
* Determine the pharmacokinetics of this drug in these patients.
* Assess the preliminary evidence of therapeutic activity of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to use of anticonvulsants known to be metabolized by the P450 hepatic enzyme complex (yes vs no).

Patients receive karenitecin IV over 60 minutes on days 1-5. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of karenitecin according to the continual reassessment method until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose associated with a dose-limiting toxicity rate of 33%.

Patients are followed every 2 months.

PROJECTED ACCRUAL: Approximately 3-24 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed anaplastic astrocytoma, anaplastic oligodendroglioma, or glioblastoma multiforme
* Progressive or recurrent disease previously treated with radiotherapy with or without chemotherapy

  * Prior low-grade disease that progressed to high-grade after therapy allowed
* Measurable disease by MRI or CT scan

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 8.5 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* Transaminases no greater than 4 times upper limit of normal

Renal:

* Creatinine no greater than 1.7 mg/dL

Other:

* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast
* No serious concurrent infection
* No other medical illness that would preclude study
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No more than 1 prior chemotherapy regimen

Endocrine therapy:

* Must be on stable dose of steroids for at least 5 days

Radiotherapy:

* See Disease Characteristics
* At least 3 months since prior radiotherapy and recovered
* No more than 1 prior course of radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent investigational agents
* At least 10 days since prior anticonvulsant drugs that induce hepatic metabolic enzymes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A. Grossman, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (8):
- United States (8):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania